CLINICAL TRIAL: NCT02024204
Title: Uncontrolled Lower Respiratory Symptoms in the World Trade Center Survivor Program
Brief Title: Uncontrolled Lower Respiratory Symptoms in the WTC Survivor Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-00448; 1U01OH010404-01A1 (NIH)
Record Dates: First submitted 2013-12-18; First posted 2013-12-31 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Lung Diseases; Medication Compliance
Keywords: World Trade Center Disaster; Environmental Exposure; Respiratory Physiology; Inflammation; Gastrointestinal Diseases; Sinus Symptoms; PTSD; Anxiety; Depression; Hypersensitivity; Spirometry; Oscillometry
MeSH Terms: conditions — Lung Diseases; Medication Adherence; Inflammation; Gastrointestinal Diseases; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Hypersensitivity | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uncontrolled LRS (Active Comparator): Patients who have uncontrolled lower respiratory symptoms (ACT < 20) at time of Visit 1 will be provided with study Advair (Fluticasone propionate 230mcg/salmeterol 21mcg) for a total of 3 months and receive medication adherence counseling Patients who have uncontrolled LRS at V1, but do not fit criteria for Step 3,4 or 5 asthma therapy according to NIH EPR III asthma guidelines will be deferred from the study until they have been seen by their physician and tried on ICS therapy.
  Interventions: Drug: Fluticasone propionate 230mcg for 3 Months; Drug: Salmeterol 21mcg for 3 Months
- Controlled LRS (Other): Patients who had symptoms at monitoring visit but are now controlled at V1 will be asked to continue their current treatment (or no treatment) and will continue with the study. They will not be provided with any medications.
  Interventions: Drug: Current Treatment or no treatment

INTERVENTIONS:
Drug: Fluticasone propionate 230mcg for 3 Months
  Other Names: Advair HFA
  Arms: Uncontrolled LRS
Drug: Current Treatment or no treatment — Patients who had symptoms at monitoring visit but are now controlled at V1 will be asked to continue their current treatment (or no treatment) and will continue with the study. They will not be provided with any medications.
  Arms: Controlled LRS
Drug: Salmeterol 21mcg for 3 Months
  Arms: Uncontrolled LRS

SUMMARY:
The purpose of this study is to understand why patients in the World Trade Center program have continuing breathing problems. This study will improve investigators understanding of breathing problems among individuals with World Trade Center exposure by allowing them to review and monitor medication use, lung function, and examine other conditions that can contribute to problems with breathing. The findings from the study will help investigators understand why some people have persistent lower respiratory symptoms (breathing problems) after their exposure to World Trade Center dust and fumes, and may help guide better management and treatment of these symptoms.

DETAILED DESCRIPTION:
Investigators will conduct a clinical study with aggressive treatment for lower respiratory symptoms in patients in the World Trade Center Environmental Health Center. Patients in the WTC EHC with uncontrolled LRS at visit 1 will be identified and placed on high-dose inhaled corticosteroids and long-acting beta agonists for three months. Adherence will be assessed at monthly visits. Patients will perform spirometry and oscillometry at baseline and after 3 months of treatment. They will also be assessed for markers of airway inflammation, bronchial hyperresponsiveness and co-morbid conditions including depression,anxiety,post-traumatic stress disorder, gastroesophageal reflux, paradoxical vocal cord motion and rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and <75
* Meet criteria for World Trade Center Environmental Health Center enrollment
* Onset of lower respiratory symptoms after 9/11/01
* Persistent lower respiratory symptoms (> 2 times per week)
* Pre-bronchodilator forced expiratory volume in one second (FEV1) within normal limits
* < 5 pack-year tobacco history
* Not current smoker
* Asthma Control Test Score ≤ 19
* Normal chest x-ray

Exclusion Criteria:

* Age < 18 years and ≥75
* Lower respiratory symptoms or asthma history pre 9/11/01
* No persistent lower respiratory symptoms
* pre-bronchodilator FEV1 within normal limits
* > 5 pack year tobacco
* Current smoker
* Abnormal Chest X-Ray or parenchymal changes on high resolution computed tomography
* Uncontrolled major chronic illness (diabetes mellitus, congestive heart failure, cancer)
* History of significant non-World Trade Center occupational or environmental exposure
* Allergy to study drug
* Pregnancy, lactation or plans to become pregnant
* Chronic oral corticosteroid use
* High risk of fatal or near-fatal asthma within the previous 2 years
* Other lung disease (Idiopathic pulmonary fibrosis,sarcoid, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Reibman, M.D, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Reibman J, Liu M, Cheng Q, Liautaud S, Rogers L, Lau S, Berger KI, Goldring RM, Marmor M, Fernandez-Beros ME, Tonorezos ES, Caplan-Shaw CE, Gonzalez J, Filner J, Walter D, Kyng K, Rom WN. Characteristics of a residential and working community with diverse exposure to World Trade Center dust, gas, and fumes. J Occup Environ Med. 2009 May;51(5):534-41. doi: 10.1097/JOM.0b013e3181a0365b. PMID 19365288
- [Background] Friedman SM, Maslow CB, Reibman J, Pillai PS, Goldring RM, Farfel MR, Stellman SD, Berger KI. Case-control study of lung function in World Trade Center Health Registry area residents and workers. Am J Respir Crit Care Med. 2011 Sep 1;184(5):582-9. doi: 10.1164/rccm.201011-1909OC. PMID 21642248

RESULTS

PARTICIPANT FLOW:
Groups:
- Visit 1 Uncontrolled LRS: Patients who have uncontrolled LRS (ACT < 20) at time of Visit 1 will be provided with study Advair (Fluticasone propionate 230mcg/salmeterol 21mcg) for a total of 3 months and receive medication adherence counseling Patients who have uncontrolled LRS at V1, but do not fit criteria for Step 3,4 or 5 asthma therapy according to NIH EPR III asthma guidelines will be deferred from the study until they have been seen by their physician and tried on ICS therapy.
  Fluticasone propionate 230mcg for 3 Months
  Salmeterol 21mcg for 3 Months
- Visit 1 Controlled LRS: Patients who had symptoms at monitoring visit but are now controlled at V1 will be asked to continue their current treatment (or no treatment) and will continue with the study. They will not be provided with any medications.
  Current Treatment or no treatment: Patients who had symptoms at monitoring visit but are now controlled at V1 will be asked to continue their current treatment (or no treatment) and will continue with the study. They will not be provided with any medications.
Period: Overall Study
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Started | 49 | 11
Completed | 49 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS | Total
Number analyzed (Participants) | 49 | 11 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [48 to 62] | 56 [47 to 62] | 56.5 [47.8 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 10 | 42
  Male | 17 | 1 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 26 | 4 | 30
  NH-White | 10 | 1 | 11
  NH-Black | 12 | 3 | 15
  Asian and Other | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 49 | 11 | 60

OUTCOME MEASURES:

1. Primary Outcome: Forced Oscillation Technique (FOT) Measures
Description: Small airway function measured pre/post BD (bronchodilator) impulse oscillometry at resistance 5 Hz (R5) and 5-20 Hz (R5-20).
Time Frame: Week 12
Measure: Median (Inter-Quartile Range); unit: resonant frequency
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
resonant frequency
  Pre BD R5 | 4.4 [3.4 to 5.7] | 3.7 [3.3 to 5.7]
  Pre BD R5-20 | 1.0 [0.5 to 1.5] | 0.6 [0.4 to 1.4]
  Post BD R5 | 4.1 [3.5 to 5.3] | 4.0 [3.4 to 5.7]
  Post BD R5-20 | 0.8 [0.4 to 1.2] | 0.6 [0.4 to 1.1]

2. Primary Outcome: Spirometry Measures
Description: Measured pre/post BD (bronchodilator). Reported as ratio: %FEV1(Liters)/FVC(Liters).
  FEV1 = forced expiratory volume at 1 second FVC = forced vital capacity
Time Frame: Week 12
Measure: Median (Inter-Quartile Range); unit: % FEV1(Liters)/FVC(Liters)
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
% FEV1(Liters)/FVC(Liters)
  Pre-BD FEV1/FVC | 78.5 [72.4 to 82.4] | 81.2 [75.3 to 83.4]
  Post-BD FEV1/FVC | 78.3 [75 to 82.2] | 77.7 [75.4 to 81.1]

3. Secondary Outcome: Number of Participants With Positive Level of Bronchial Hyperreactivity (BHR)
Description: To test whether bronchial Hyperreactivity (BHR), assessed by methacholine challenge, is associated with uncontrolled lower respiratory symptoms.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
Participants | 18 | 6

4. Secondary Outcome: Number of Participants With Positive Level of Paradoxical Vocal Fold Movement (PVFM)
Description: measured by laryngoscopic visualization at rest or after provocation with various odors or exercise.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
Participants | 21 | 6

5. Secondary Outcome: Total IgE (Immunoglobulin E) Levels
Description: IgE levels were obtained by blood test - the total amount of blood drawn is 30 mL.
Time Frame: Week 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
ng/mL | 41 [20 to 135] | 31 [21.5 to 57]

6. Secondary Outcome: Total EoS (Eosinophil) Counts
Description: EoS counts were obtained by blood test - the total amount of blood drawn is 30 mL.
Time Frame: Week 1
Measure: Median (Inter-Quartile Range); unit: eosiniphils *10^9/Liter
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
eosiniphils *10^9/Liter | .10 [.10 to .20] | .10 [.10 to .10]

7. Secondary Outcome: Levels of Fractional Exhaled Nitric Oxide (FeNO)
Description: Measured using a portable device that measures the level of nitric oxide in parts per billion (PPB) in the air slowly exhaled out of the patient's lungs.
Time Frame: Week 12
Measure: Median (Inter-Quartile Range); unit: parts per billion (ppb)
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
parts per billion (ppb) | 17.8 [14 to 22.2] | 13 [10.2 to 13.9]

8. Secondary Outcome: Score on Voice Handicap Index 10 (VHI-10)
Description: Voice Handicap Index 10 is a measure of laryngeal dysfunction or hypersensitivity to capture the "overall" state of voice handicap. The normative value for this instrument is 2.83, with a score > 11 considered abnormal. There are 10 statements that are scored between 0 and 4 (0= never, 4= always). The total range is 0-40, where 40 is highest level of dysfunction.
Time Frame: Week 12
Measure: Median (Inter-Quartile Range); unit: score on VHI-10 scale
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
score on VHI-10 scale | 7 [1 to 17] | 1 [0.0 to 9.8]

9. Secondary Outcome: Rhinosinusitis Score on International Classification of Sleep Disorders (ICSD)
Description: For rhinosinusitis symptoms, the ICSD scoring system was used, with a likert scale of 1-10 for each symptom (total range of scale = 1-60, with higher scores reflecting more symptoms).
Time Frame: Week 12
Measure: Median (Inter-Quartile Range); unit: score on ICSD scale
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
score on ICSD scale | 35 [24 to 42.5] | 26 [18.2 to 29.5]

10. Secondary Outcome: Score on Leicester Cough Questionnaire (LCQ)
Description: For rhinosinusitis symptoms, the Leicester Cough Questionnaire (LCQ) was used - a cough-specific health status questionnaire that assesses the physical, psychological, and social domains of cough. The LCQ is made up of 19 items; the total score range is 3-21; a higher score is associated with better health.
Time Frame: Week 12
Measure: Median (Inter-Quartile Range); unit: score on LCQ scale
Arm/Group | Visit 1 Uncontrolled LRS | Visit 1 Controlled LRS
Number analyzed (Participants) | 49 | 11
score on LCQ scale | 12 [8.9 to 15.4] | 15.6 [12.7 to 20.2]

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Uncontrolled LRS: Patients who have uncontrolled lower respiratory symptoms (ACT < 20) at time of Visit 1 will be provided with study Advair (Fluticasone propionate 230mcg/salmeterol 21mcg) for a total of 3 months and receive medication adherence counseling Patients who have uncontrolled LRS at V1, but do not fit criteria for Step 3,4 or 5 asthma therapy according to NIH EPR III asthma guidelines will be deferred from the study until they have been seen by their physician and tried on ICS therapy.
  Fluticasone propionate 230mcg for 3 Months
  Salmeterol 21mcg for 3 Months
Arm/Group | Uncontrolled LRS | Controlled LRS
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/11
Other Adverse Events (participants affected / at risk) | 0/49 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT02024204/Prot_SAP_000.pdf